CLINICAL TRIAL: NCT05346952
Title: A Phase 3，Randomized，Open，Parallel Controlled, Multi-center Study of TQB2450 Injection Plus Chemotherapy Followed by TQB2450 Plus Anlotinib Versus Tislelizumab Plus Chemotherapy Followed by Tislelizumab as a First-line Treatment on Patient With Advanced Non-squamous NSCLC
Brief Title: A Study of TQB2450 Injection Plus Chemotherapy Followed by TQB2450 Plus Anlotinib Versus Tislelizumab Plus Chemotherapy Followed by Tislelizumab in the Treatment of First-line Non-squamous Non-small Cell Lung Cancer(NSCLC).
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-Ⅲ-11
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Advanced Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450 injection + carboplatin + pemetrexed (Experimental): TQB2450 injection：1200 mg, Intravenous drip d1； carboplatin ：Area Under Curve 5mg/mL/min，Intravenous drip d1；Pemetrexed: 500mg/m2，Intravenous drip d1.The above schemes are repeated every three weeks. After 4 cycles, the regimen is changed to TQB2450 injection（1200 mg, Intravenous drip d1）+Pemetrexed（500mg/m2，Intravenous drip d1）+ Anlotinib (10mg, peros every day, d1-14) . The regimen is repeated every 3 weeks until the disease progresses.
  Interventions: Drug: TQB2450 injection, Tilelizumab injection, Anlotinib hydrochloride capsule, Pemetrexed disodium injection, Carboplatin injection
- TQB2450 injection + Anlotinib + Pemetrexed (Active Comparator): Tilelizumab: 200 mg, Intravenous drip d1;carboplatin : AUC 5mg/mL/min, Intravenous drip d1；Pemetrexed: 500mg/m2, Intravenous drip d1.The above schemes are repeated every three weeks. After 4 cycles, the regimen is changed to Tilelizumab (200 mg, Intravenous drip d1)+Pemetrexed (500mg/m2，Intravenous drip d1).The regimen is repeated every 3 weeks until the disease progresses.
  Interventions: Drug: TQB2450 injection, Tilelizumab injection, Anlotinib hydrochloride capsule, Pemetrexed disodium injection, Carboplatin injection

INTERVENTIONS:
Drug: TQB2450 injection, Tilelizumab injection, Anlotinib hydrochloride capsule, Pemetrexed disodium injection, Carboplatin injection — PD-L1(programmed cell death-Ligand 1) may be expressed on tumor cells and/or tumor-infiltrating immune cells, which can inhibit the anti-tumor immune response in the tumor microenvironment. On T cells and antigen-presenting cells, PD-L1 binding to PD-1 (programmed cell death-1) and B7.1 receptors inhibits cytotoxic T cell activation, T cell proliferation, and cytokine production.

SUMMARY:
This is Phase 3, randomized, open-label, parallel controlled study designed to compare the efficacy and safety of TQB2450 in combination with platinum-containing chemotherapy followed by TQB2450 plus Anlotinib versus tislelizumab in combination with platinum-containing chemotherapy followed by tislelizumab in locally advanced (stage ⅢB/ⅢC), metastatic or recurrent ( Stage IV) non-squamous NSCLC cancer. The primary endpoint is Progression Free Survival (PFS) assessed by IRC.

ELIGIBILITY:
Inclusion Criteria:

* 1 According to the 8th edition of the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification, the TNM staging of lung cancer is locally advanced (stage ⅢB/ⅢC), metastatic or recurrent ( Stage IV) NSCLC patients.
* 2 Between the ages of 18-75 years (calculated based on the date of signing ICF); male or female; Eastern cooperative oncology group (ECOG) score 0-1; estimated survival time ≥ 3 months.
* 3 According to the RECIST 1.1 standard, there is at least one measurable lesion. If the measurable lesion is located in the radiotherapy area, it should be clearly defined as a progressive state.
* 4 Patients who have not received systemic anti-tumor therapy for advanced, recurrent or metastatic diseases in the past. For those who have received adjuvant chemotherapy in the past, the interval between the recurrence time and the last adjuvant chemotherapy should be at least 6 months; The interval between the end of previous radiotherapy for chest and this treatment should be more than 6 months, and the interval between palliative radiotherapy for chest and this treatment should be more than 7 days.
* 5 Tumor tissue sections that have not undergone radiotherapy at or after the diagnosis of advanced or metastatic NSCLC must be provided. Tumor tissue samples must be archived samples or freshly obtained samples within 12 months before randomization.
* 6 For non-squamous NSCLC, patients with no EGFR sensitive mutations, ALK fusion, ROS1 fusion
* 7 The function of main organs are well and meet the following standards:
* 8 a. Routine blood examination standards (without blood transfusion or correction with hematopoietic stimulating factor drugs within 14 days before screening): i. Absolute neutrophil count (ANC) ≥1.5×109 /L; ii. Platelets ≥100×109 /L; iii. Hemoglobin ≥90 g/L. b. The blood biochemical examination shall meet the following standards: i. Total bilirubin (TBIL) ≤ 2 × upper limit of normal (ULN) (Patients with Gilbert syndrome ≤ 3 × ULN); ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5×ULN. If it is accompanied by liver metastasis, ALT and AST≤5×ULN; 8.iii. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance estimated by Cockcroft-Gault glomerular filtration formula ≥60 mL/min; iv. Serum albumin (ALB) ≥30g/L. c. Urine routine examination standard: urine routine indicates urine protein <++; if urine protein ≥++, it is necessary to confirm that the 24-hour urine protein quantitative ≤1.0 g.

  d. Blood coagulation test standards: prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR)≤1.5×ULN (no anticoagulant therapy).

  e. Thyroid Stimulating Hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be examined. If T3 and T4 levels are normal, it can be selected.

  f. Heart color Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.

  g. 12-lead ECG evaluation: QTc<450ms (male), QTc<470ms (female).
* 9 Women of childbearing age should agree to use effective contraceptive measures during the study period and 6 months after the end of the study, and have a negative serum pregnancy test within 7 days before the study enrollment; men should agree to the study period and 6 months after the end of the study period Effective contraceptive measures must be used internally.
* 10 The subjects voluntarily joined the study, signed the informed consent form, and had good compliance.

Exclusion Criteria:

* 1 Tumor disease and medical history:

  1. Brain metastases without local treatment; Note: Subjects who have previously received brain metastasis therapy and meet all the following criteria can participate in this study: i. Only supratentorial and cerebellar metastases; ii. The condition needs to be stable for ≥4 weeks and no new brain metastases or brain metastases are found Expanded imaging evidence; iii. The subject must have stopped corticosteroids/dehydrator for at least 2 weeks before starting to use the trial drug;
  2. There are midbrain, pons, medulla oblongata, spinal cord and meningeal metastases；
  3. Other malignant tumors appeared or were present within 3 years. The following two cases can be included: other malignant tumors treated by single operation have achieved 5-year Disease-free survival (DFS) in a row; The cured cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [ta (non-invasive tumor), tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
  4. Central type, cavity squamous cell carcinoma (primarily in the main bronchus and around the hilar);Imaging shows that the tumor invades large blood vessels or is unclearly separated from the blood vessels, or the investigator judges that the tumor is likely to invade important blood vessels and cause fatal bleeding during the subsequent study(The major vessels in the chest include pulmonary aorta, left pulmonary artery, right pulmonary artery, four pulmonary veins, superior vena cava, inferior vena cava and aorta);
  5. Severe bone injury caused by tumor bone metastasis, including pathological fracture of weight-bearing bone and spinal cord compression that occurred within 6 months or is expected to occur in the near future(Such as spine, pelvis, femur, tibia, phalanges, calcaneus, etc.);
  6. Patients with serous cavity (thoracic cavity, abdominal cavity, or pericardial cavity) that require repeated drainage to relieve clinical symptoms (as determined by the investigator), or who have received drainage of serous cavity effusion for the purpose of treatment within 2 weeks before treatment.
* 2 Previous anti-tumor treatments:

  1. Received the treatment of proprietary Chinese medicines with anti-tumor indications specified in the NMPA approved drug instructions within 2 weeks before the start of the study treatment(Including compound cantharidin capsules, Kangai injection, Kanglaite capsule/injection, Aidi injection, brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, Huachansu capsule, etc.);
  2. Previously received related immunotherapy drugs for programmed death 1 (PD-1), PD-L1, cytolytic T lymphocyte-associated antigen-4 (CTLA-4), etc.;
  3. Previous use of anti-angiogenic drugs such as bevacizumab, anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, regorafenib, fruquintinib, etc.;
  4. Patients who have been vaccinated with immunomodulatory drugs within 30 days before starting treatment(Such as interleukin-2, thymosin, lentinan, etc.);
  5. Failure to recover from the toxicity and/or complications of previous interventions to CTCAE ≤1, except for hair loss and peripheral neuropathy ≤2;
* 3 Combined diseases and medical history:

  1. Liver cirrhosis, active hepatitis*;(Note: active hepatitis (hepatitis B reference: HBV-DNA > 1*103 copy /mL or > 2000IU/mL) when HBsAg is positive. Hepatitis C reference: HCV antibody is positive, and HCV titer detection value exceeds the upper limit of normal value);
  2. Renal abnormalities: i.Renal failure requires hemodialysis or peritoneal dialysis; ii.Previous or existing nephrotic syndrome, chronic nephritis.
  3. Cardiovascular and cerebrovascular abnormalities： i.Patients with previous or present heart failure, degree II or above heart block: ii.Myocardial infarction or unstable angina, supraventricular or ventricular arrhythmia with clinical significance need treatment or intervention; iii.Vascular embolism and cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage and cerebral infarction) occurred within 9 months（ Prophylactic use of anticoagulant therapy is allowed for patients with thrombotic tendency or undergoing anticoagulant therapy.) iv.After more than two kinds of drug treatment, blood pressure control is still not ideal (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg).
  4. Gastrointestinal abnormalities: i.Inability to take medications (such as inability to swallow, intestinal obstruction, etc.); ii.A history of malabsorption syndrome or other diseases that interfere with gastrointestinal absorption; iii.Received treatment for active peptic ulcer in the past 6 months; iv.Despite the maximum medical treatment, chronic diarrhea of grade 2 and above continues to occur; v.Other conditions determined by the researcher that may cause gastrointestinal bleeding and perforation.
  5. History of immunodeficiency:

  i.Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases; ii.Active autoimmune disease or history of autoimmune disease, including but not limited to Crohn's disease, ulcerative colitis, autoimmune hepatitis/enteritis/vasculitis/nephritis, etc.

iii.Prepare to undergo or have previously received an organ transplant; iv.Patients who require systemic or topical immunosuppressive therapy to achieve immunosuppressive purposes and need to continue to use them within two weeks before randomization (except for glucocorticoid daily dose <10 mg prednisone or other equivalent hormones).

Note: Hormone replacement therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered as systemic therapy and allowed to be used.

f. Bleeding risk: i.Suffered from bleeding or coagulopathy within 28 days before the start of treatment or was using warfarin, aspirin and other antiplatelet agglutination drugs (except for aspirin ≤100 mg/d preventive drugs); ii.Had hemoptysis >2.5 mL/day in 28 days before the start of treatment; iii.Regardless of the severity, patients with any history of bleeding or coagulopathy; iv.Received major surgical treatment, open biopsy, etc. within 28 days before the start of the study treatment; v.Long-term unhealed wounds or fractures, except for pathological fractures; g. Poor control of type I diabetes or II diabetes (fasting blood glucose (FBG)> 10mmol/L); h. Severe infections within 4 weeks before the start of study treatment, including but not limited to hospitalization due to bacteremia, severe pneumonia, or other severe infections; subjects with ≥ grade 2 active infections within 4 weeks before the start of study treatment Or fever of unknown cause occurred during the screening period and before the first administration>38.0℃; i. Past or existing pneumoconiosis, interstitial pneumonia, (non-infectious) pneumonia that requires adrenal corticosteroid therapy, currently suffering from other types of pneumonia ≥2, or lung function tests confirmed severely impaired lung function (Forced Expiratory Volume in the first second (FEV1) or diffusing capacity of lung for carbon monoxide(DLCO) or DLCO per alveolar volume (DLCO /VA) accounts for the expected value %<40%) and other objective evidence; j. Patients with active tuberculosis within 1 year before enrollment; subjects with a history of active pulmonary tuberculosis infection 1 year ago must provide clear evidence of cure before enrollment; if tuberculosis is suspected during the screening period, chest radiographs and sputum must be passed Enter the group only after the liquid and clinical symptoms are eliminated; k. Allergies, or a history of severe allergies in the past, or severe hypersensitivity reactions after receiving other monoclonal antibody treatments, or known allergies to the ingredients of the study drug excipients; l. Previous history of severe mental disorders; m. People with a history of drug abuse, alcohol or drug abuse;

* 4 The end of the previous clinical study (last dose) is less than 4 weeks or the study drug's 5 half-lives, whichever is shorter.
* 5 Live attenuated vaccine vaccination history within 28 days before randomization or planned live attenuated vaccination during the study period. Seasonal influenza vaccine for injection is usually an inactivated virus vaccine and is allowed to be vaccinated during the study period.
* 6 Female patients during pregnancy or lactation.
* 7 According to the investigator's point of view, it may increase the risks associated with participating in the study, or other severe, acute or chronic medical diseases or laboratory abnormalities that may interfere with the interpretation of the study results, or other reasons that are not suitable for participating in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by IRC | Up to 2 years
  The period from the first use of the drug to disease progression or death (whichever occurs first).
Overall survival (OS) | Up to 3 years
  Time from randomization to death
According to response evaluation criteria in solid tumours 1.1（RECIST1.1）standard and iRECIST （Immune-related response evaluation criteria in solid tumours ）standard researcher's assessment of progression-free survival (PFS) | Up to 2 years
  The period from the first use of the drug to disease progression or death (whichever occurs first).
Objective Response Rate (ORR) | Up to 2 years
  Proportion of patients whose tumor volume shrinks to a predetermined value and maintains the minimum time limit
Disease Control Rate (DCR） | Up to 2 years
  Proportion of subjects whose tumors shrink or remain stable for a certain period, including CR, PR and stable disease SD
Duration of Remission (DOR) | Up to 2 years
  The period from firstly-recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurs first) .
TTR | Up to 2 years
  Time from randomization to onset of remission (PR)

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)，as well as abnormal laboratory examination indicators. | Up to 2 years
  The proportion of AEs and SAEs recorded afte signing the informed consent form(ICF).

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality, China